CLINICAL TRIAL: NCT03908255
Title: Impact of Branched-chain Amino Acid Supplementation on Quality of Life and Overall Survival in Patients Receiving Liver Directed Therapy for Hepatocellular Carcinoma
Brief Title: Branched-chain Amino Acid Supplementation for Hepatocellular Carcinoma
Acronym: BCAA in HCC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dr. Marshall left UMC and LSU Health Sciences Center.
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: University Medical Center-New Orleans (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BCAA in HCC Intervention
Record Dates: First submitted 2018-12-07; First posted 2019-04-09 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-08

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis; Liver Failure
Keywords: branch chain amino acid; nutritional supplement; malnutrition; decompensated liver failure
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Liver Failure; Malnutrition | interventions — Amino Acids; maltodextrin

STUDY DESIGN:
Intervention Model Description: This study design will be a double-blinded, randomized clinical control trial in which treatment-naïve patients diagnosed with HCC will be screened at baseline before being randomized to either a treatment group, which will receive standard of care and BCAA supplement, or to a control group which will receive standard of care and a maltodextrin placebo. Both groups will receive liver directed therapy including transarterial chemoembolization (TACE) at baseline. In the intervention group, patients will receive current standard of care and consume BCAA supplements beginning two weeks prior to liver directed therapy and continue supplementation for the following 12 months. The control group will receive current standard of care, consume a maltodextrin placebo beginning two weeks prior to liver directed therapy and continue supplementation for the following 12 months.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will receive current standard of care (locoregional therapy of the liver, serial bloodwork and imaging, serial assessments in clinic), consume a maltodextrin placebo supplement beginning two weeks prior to liver directed therapy and continue supplementation for the following 12 months.
  Interventions: Other: maltodextrin
- Intervention Group (Experimental): In the intervention group, patients will receive current standard of care (locoregional therapy of the liver, serial bloodwork and imaging, serial assessments in clinic) and consume BCAA supplements beginning two weeks prior to liver directed therapy and continue supplementation for the following 12 months.
  Interventions: Drug: Branch Chain Amino Acid

INTERVENTIONS:
Drug: Branch Chain Amino Acid — Nutritional supplementation
  Other Names: Do Vitamins BCAA
  Arms: Intervention Group
Other: maltodextrin — Placebo
  Arms: Control Group

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cause of cancer death among men. While several new treatment options have recently become available, they are costly and have a potential for significant, adverse side effects. Many patients diagnosed with HCC also suffer from underlying liver disease, including cirrhosis. As many as 80-90% of patients diagnosed with HCC also have cirrhosis. Protein-energy malnutrition (PEM) in cirrhosis is as high as 65-90% and significantly increases the risk of morbidity and mortality as well as decreased quality of life.

Branched-chain amino acid (BCAA) supplementation has been extensively studied for usefulness in liver disease, specifically to treat hepatic encephalopathy to and preserve and restore muscle mass. Maintenance of liver function and prevention of PEM are essential for improving outcomes in patients with HCC. Branched-chain amino acid supplementation in HCC has been studied extensively in China & Japan with multiple studies showing improvements in liver function, progression-free survival, and overall survival. Additionally, patients in treatment groups have shown improvement in quality of life indicators. However, these results have yet to be replicated in the United States. Branched-chain amino acid supplementation may be a safe, low-cost approach to improve survival, liver function indicators, and quality of life for patients diagnosed with HCC.

In this study, patients with primary HCC will be randomized to either a treatment group, which will receive standard of care and BCAA supplement or to a control group which will receive standard of care and a maltodextrin placebo. Both groups will receive liver-directed therapy including transarterial chemoembolization (TACE) and thermal ablation. All patients will complete a quality of life survey (FACT-Hep) at each visit.

DETAILED DESCRIPTION:
Products or Devices to be Studied:

Branched Chain Amino Acid anhydrous blend (1250mg valine, 2500mg leucine, 1250mg isoleucine) Pre-assigned IND number: 140871 Holder of the IND (Richard Marshall, MD)

Purpose of the Study:

Aim: To evaluate the effect of branched-chain amino acid (BCAA) supplementation on progression-free survival and overall survival in patients diagnosed with hepatocellular carcinoma (HCC).

Rationale:

Hepatocellular carcinoma (HCC) is the most common adenocarcinoma affecting the liver. Approximately 14 million people are affected globally and the number of cases is expected to increase to 22 million by 2032. In the United States, HCC accounts for 5% of all cancer-related deaths and has a 1-year survival rate of 41.5% and a 5-year survival rate of 16.5%. Although several new treatment options have recently become available, they are expensive and show a strong potential for adverse side effects. Regardless of treatment modality, liver function maintenance is an essential component for improving outcomes in patients with HCC.

The liver functions as a primary site for macronutrient, enzyme, vitamin, bile acid, and heme metabolism as well as the breakdown and excretion of toxic waste products of metabolism. Among the liver's many roles is the production of albumin, a serum protein responsible for maintaining oncotic pressure and the transportation of nutrients throughout the body. Low levels of albumin (hypoalbuminemia) are associated with severe malnutrition and can lead edema due to decreased oncotic pressure. Hepatic tissue damage, tumor formation, and tumor proliferation decreases the liver's functional capacity for executing these processes.

Chronic injury to the hepatocytes can lead to the development of hepatocellular carcinoma. Once developed, tumor cells and stromal cells form a network called the tumor microenvironment which further contributes to tumor proliferation. Treatments to disrupt the microenvironment (e.g. sorafenib) may be successful in reducing fibrosis, liver damage, inflammation, and angiogenesis. These treatments are not without serious side effects including: myocardial infarction, bleeding problems, bowel perforation, and hypertension to name a few.

Therapeutic approaches to manage symptoms associated with HCC include late evening snacks and protein supplementation. The rationale purports that improvements in nutritional quality will alleviate catabolic stress, thereby reducing risks of associated complications of malnutrition including: protein energy malnutrition, hypoalbuminemia, and hepatic encephalopathy. Further, the branched-chain amino acids (BCAA) valine, leucine, and isoleucine may act on the same signaling pathways of chemotherapeutic pharmaceuticals in addition to improving nutritional status in patients with HCC.

Recently, BCAA supplementation has been explored as a possible treatment for hepatocellular carcinoma in conjunction with standard of care in Japan and China. A recent meta-analysis of clinical studies from China and Japan supports the safety of BCAA supplementation and the possible benefit of improving liver functional reserves and quality of life. However, significant differences in study designs and BCAA doses make inferring conclusions from these studies difficult. Moreover, studies don't adequately control for differences in dietary intake between treatment groups which may skew results. To date, no clinical trials have been conducted in the United States that examine the effects of BCAA supplementation in patients with HCC. The purpose of this study is to examine the safety, efficacy, and feasibility of BCAA supplementation in patients with HCC who undergo locoregional therapies.

Study Procedures:

Current standard of care for hepatocellular carcinoma consists of physician monitoring following liver directed therapy and does not include any nutrition or dietary intervention beyond meeting basic nutritional needs. The study procedures differ from standard of care only by the addition of either a BCAA supplement or maltodextrin placebo, administration of a quality of life survey (FACT-Hep), and a personalized diet prescription.

To ensure protein and energy intake is equivalent between groups, individualized diets will be calculated by the dietitian based on current height, weight, and stress factors for those in both arms of the study. The corresponding meal plan will be administered by the research pharmacist. The intervention group receiving 10g of BCAA daily will receive a meal plan that reflects a protein deficit of 10g below estimated needs (which will be covered by the BCAA supplement).

Subjects:

Forty subjects will be enrolled. Patients who are seeking treatment in the interventional radiology department at University Medical Center (UMC) will comprise the sample.

Duration of the Study:

Enrollment of the full sample will take approximately 36 months and each participant will be followed for 12 months after enrollment and initiation of the treatment. This study would conclude approximately 48 months following first enrollment. Each individual's participation in the study will be 12-14 months following their enrollment.

Implementation Summary:

Patients will be educated about the study by an interventional radiologist and oncology dietitian during their first visit to the interventional radiology clinic at UMC. After providing informed consent to participate in the study, patients will be immediately started on their dietary supplement (BCAA or placebo) for two weeks. BCAA supplements will be dispensed a UMC pharmacist. Patients will then have a brief hospital stay at UMC (typically ranging 6-24 hours) to receive their TACE and/or ablation procedure. All patients will be assessed by an interventional radiologist or nurse practitioner prior to discharge, and those undergoing a TACE procedure will also have a comprehensive metabolic panel (CMP) drawn. After discharge patients will have a one month, three month, 6 month, 9 month, and 12 month follow up in the interventional radiology clinic where they will meet with the physician and dietitian. A detailed list of procedures is provided below. Patients may require additional visits if it is determined that they need additional local therapies (repeat TACE and/or Ablation).

Risks of Interventions:

Branched-chain amino acid supplementation. Risks: Based on data from prior studies, participants receiving BCAA supplementation protocol may experience nausea, vomiting, abdominal pain, diarrhea or hypertension.

Maltodextrin supplementation. Risks: Maltodextrin is a sugar. Consuming maltodextrin may cause a temporary rise in blood sugar. However the amounts consumed for this study will be very small. There are no known risks associated with its use. Maltodextrin is affirmed by the FDA as GRAS per Title 21 of the Code of Federal Regulations Section 184.1444.

Fact-Hep questionnaire. Risks: there are no known risks to questioning about health-related quality of life.

Data Safety Monitoring:

Definition:

Serious adverse event (SAE): events including death, a life-threatening adverse experience, inpatient hospitalization, prolongation of existing hospitalization, and persistent or significant disability or incapacity.

Adverse event (AE): any health-related, unfavorable or unintended medical occurrence that happens throughout study participation. Examples of adverse events include but are not limited to the following:

A clinically significant laboratory or clinical test result. An event that results in missing a study visit. An event that requires a visit to a physician. An event that occurs as a result of a study procedure. Unanticipated or untoward medical events that may be study related.

Monitoring Plan:

Adverse events will be reported to the principal investigator as they are collected from the participant. Adverse event data will be analyzed quarterly, whereas serious or life-threatening adverse events will necessitate immediate reporting and follow-up. It is anticipated that most adverse events will be mild and the participant will be able to resume activities within one to two days of reporting the event.

SAEs that are unanticipated, serious, and possibly related to the study intervention will be reported to the IRB and FDA. Unexpected problems involving risks to participants or others include incidents only if the incident is unexpected, related or possibly related to participation in the research, and indicated that subjects or others are at a greater risk of harm than was previously known or recognized. A SAE will result in the unblinding of the participant and will be reported to the IRB and FDA per CFR § 312.32(c)(5). Any action resulting in unblinding, and/or a temporary or permanent suspension of this study (e.g., IRB actions, or actions by the PI and/or co-investigators) will be reported to the appropriate officials.

Aggregate comparisons of AE and SAE between study arms will occur after 50% of the participants are enrolled. If there is evidence of a significant, clinically relevant difference in SAE between groups, the study will be unblinded; and in the event the BCAA group experiences significantly fewer SAEs, the placebo group will be offered the BCAA supplement. Conversely, if the BCAA group experiences significantly more SAEs, the supplementation will be terminated and follow-up will continue as planned.

Statistical Analysis:

A total of 40 subjects will be recruited (20 in each intervention and control group). Sample size was determined to achieve a power of 0.8 for a two-sided test (α = 0.05) for a balanced study design. The results of the power analysis indicate that this can be achieved with a sample ranging from 13-21 patients in each arm with the assumption that 1 year mortality will be 41.5% in the control group (mortality rate derived from epidemiological data) and a mortality rate ranging from 85 - 95% in the intervention group. Progression-free survival and overall survival will be examined using survival regression analyses while controlling for relevant covariates (age, demographics, etc.). Quality of life, Child Pugh score, and biomarkers of liver function will be examined using repeated measures ANOVA with contrasts between the treatment groups. Tolerability of the BCAA supplement will be assessed by examining the number of adverse effects reported by participants. The severity of the adverse events will be assessed by the physician and frequency differences between groups will be compared using Χ² test statistic.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with HCC and deemed a candidate for nonsurgical local therapy (TACE and/or percutaneous ablation)
* Have a Child-Pugh score < 6
* Are at least 18 years of age or older
* Otherwise healthy adults
* Provide written consent to participate

Exclusion Criteria:

* Have a diagnosis of renal failure
* Have a Child-Pugh score > 6
* Consume > 60g alcohol intake per day
* Have been diagnosed with branched-chain ketoaciduria (maple syrup urine disease)
* Have hepatic encephalopathy
* Have been diagnosed with a medical condition that warrants a low-protein diet
* Are currently taking insulin or metformin
* Pregnant women
* Younger than 18 years of age
* Are unable to provide consent
* Are incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 24 months after enrollment
  Overall survival after after Day 0 of study (date of HCC treatment)

SECONDARY OUTCOMES:
Tolerability and Use of BCAA Supplement: use of the supplement as greater than 50% compliance or less than 50% compliance | At every clinic visit up to 24 months after enrollment
  Assess the supplement's tolerability and adherence to branched chain amino acid supplementation schedule by evaluating use of the supplement as greater than 50% compliance or less than 50% compliance.
Progression Free Survival | Up to 24 months after enrollment
  Growth or metastasis of HCC measured in days after Day 0 of study (date of HCC treatment) using Liver Imaging Reporting and Data System (LI-RADS) 2018 "Threshold growth", "Tumor Viability" criteria (per the American College of Radiology (ACR), https://www.acr.org/-/media/ACR/Files/RADS/LI-RADS/LI-RADS-2018-Core.pdf?la=en)as well as RECIST 1.1 criteria (per the RECIST Working Group, http://recist.eortc.org/recist-1-1-2/)
Event Free Survival | Up to 24 months after enrollment
  Evaluate event free survival in days after Day 0 of study (date of HCC treatment). Events include tumor growth, metastasis, portal vein thrombosis, jaundice, hepatic encephalopathy, new onset or worsening ascites, bleeding diathesis requiring admission, death, hospital admission related to liver disease or hepatocellular carcinoma, allergic reaction to supplement or placebo, other disease related to supplement, placebo, hepatocellular carcinoma or advanced liver disease.
Quality of life using FACT-Hep | Every 6 months up to 24 months after enrollment
  Quality of life will be measured objectively by through use of the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT Hep), version 4, Questionnaire. This is a 46 question survey that will be given to participants every 6 months to determine their overall quality of life. Participants answer questions related to symptoms experienced in the last 7 days by circling responses that include "Not at all" (0), "A little bit" (1), "Somewhat" (2), "Quite a bit" (3), "Very much" (4) and the numerical score is used to calculate a total score. Higher scores are associated with higher quality of life. Subcategories exist and numerical totals for subcategories (including physical well being, social/family well being, emotional well being, functional well being, and additional concerns) will be used to score specific characteristics. A link is attached as a reference.

OTHER OUTCOMES:
Child Pugh Score | At every clinic visit up to 24 months after enrollment
  The Child Pugh Score, used to measure overall liver health and prognosis of liver disease, will be calculated (after each lab measurement and clinical assessment using serum albumin, bilirubin, international normalized ratio, presence and severity of ascites and presence and severity of hepatic encephalopathy will be assessed using a numeric score assigned to each category. Total scores are a sum of each category and a higher total is associated with a worse prognosis. No subclassifications will be applied. Please see the reference section for a clinical application of this scale.
Weight | At every clinic visit up to 24 months after enrollment
  Measurement of weight in both kilograms and pounds
Height | Every 3 months up to 24 months after enrollment
  Height will be measured in inches, centimeters or meters and converted using conversion factors to inches, centimeters or meters at each clinic visit
Body mass index | Every 3 months up to 24 months after enrollment
  Weight and height will be combined to report BMI in kg/m^2
Aspartate aminotransferase | Every 3 months up to 24 months after enrollment
  Serum aspartate aminotransferase in units per liter
Alanine aminotransferase | Every 3 months up to 24 months after enrollment
  Serum alanine aminotransferase in units per liter
Alkaline phosphatase | Every 3 months up to 24 months after enrollment
  Serum alkaline phosphatase in units per liter
Albumin | Every 3 months up to 24 months after enrollment
  Serum albumin measurement in grams per deciliter
Bilirubin | Every 3 months up to 24 months after enrollment
  Serum bilirubin measurement in milligrams per deciliter
Platelet count | Every 3 months up to 24 months after enrollment
  Serum platelet count in thousands per microliter
International normalized ratio (INR) | Every 3 months up to 24 months after enrollment
  Measurement of coagulation (unitless)

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Marshall, MD, Principal Investigator — Louisiana State University Health Sciences Center
Locations (1):
- University Medical Center New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared in collaboration with the current investigators for future studies in which branched chain amino acids for treatment of liver disease are studied in a similar manner to this protocol. All collected data may be made available after local Institutional Review Board authorization, de-identification through a secure method of data transfer (encrypted file sharing) and kept on a secure server.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The time frame for data sharing will begin after initial publication and will extend for 5 years.
  After this point, data will be purged from secured servers and will no longer be available for sharing.
Access Criteria: A request for data will be made through the principal investigator of this study, who is responsible for data storage. Requests will be made to local Institutional Review Boards prior to de-identified data release.

REFERENCES:
- [Result] Takeda H, Nishikawa H, Iguchi E, Ohara Y, Sakamoto A, Saito S, Nishijima N, Nasu A, Komekado H, Kita R, Kimura T, Osaki Y. Effect of treatment with branched-chain amino acids during sorafenib therapy for unresectable hepatocellular carcinoma. Hepatol Res. 2014 Mar;44(3):302-12. doi: 10.1111/hepr.12125. Epub 2013 Apr 29. PMID 23607614
- [Result] Nojiri S, Fujiwara K, Shinkai N, Iio E, Joh T. Effects of branched-chain amino acid supplementation after radiofrequency ablation for hepatocellular carcinoma: A randomized trial. Nutrition. 2017 Jan;33:20-27. doi: 10.1016/j.nut.2016.07.013. Epub 2016 Aug 8. PMID 27908546
- [Result] Imanaka K, Ohkawa K, Tatsumi T, Katayama K, Inoue A, Imai Y, Oshita M, Iio S, Mita E, Fukui H, Yamada A, Nakanishi F, Inada M, Doi Y, Suzuki K, Kaneko A, Marubashi S, Ito Y, Fukui K, Sakamori R, Yakushijin T, Hiramatsu N, Hayashi N, Takehara T; Osaka Liver Forum. Impact of branched-chain amino acid supplementation on survival in patients with advanced hepatocellular carcinoma treated with sorafenib: A multicenter retrospective cohort study. Hepatol Res. 2016 Sep;46(10):1002-10. doi: 10.1111/hepr.12640. Epub 2016 Jan 26. PMID 26690886
- [Result] Chen L, Chen Y, Wang X, Li H, Zhang H, Gong J, Shen S, Yin W, Hu H. Efficacy and safety of oral branched-chain amino acid supplementation in patients undergoing interventions for hepatocellular carcinoma: a meta-analysis. Nutr J. 2015 Jul 9;14:67. doi: 10.1186/s12937-015-0056-6. PMID 26155840
- [Result] Au KP, Chan SC, Chok KS, Chan AC, Cheung TT, Ng KK, Lo CM. Child-Pugh Parameters and Platelet Count as an Alternative to ICG Test for Assessing Liver Function for Major Hepatectomy. HPB Surg. 2017;2017:2948030. doi: 10.1155/2017/2948030. Epub 2017 Aug 29. PMID 28951631
- [Result] Chernyak V, Fowler KJ, Kamaya A, Kielar AZ, Elsayes KM, Bashir MR, Kono Y, Do RK, Mitchell DG, Singal AG, Tang A, Sirlin CB. Liver Imaging Reporting and Data System (LI-RADS) Version 2018: Imaging of Hepatocellular Carcinoma in At-Risk Patients. Radiology. 2018 Dec;289(3):816-830. doi: 10.1148/radiol.2018181494. Epub 2018 Sep 25. PMID 30251931
- [Result] Gmur A, Kolly P, Knopfli M, Dufour JF. FACT-Hep increases the accuracy of survival prediction in HCC patients when added to ECOG Performance Status. Liver Int. 2018 Aug;38(8):1468-1474. doi: 10.1111/liv.13711. Epub 2018 Feb 20. PMID 29389088
- See also: LI-RADS v2018 — https://www.acr.org/-/media/ACR/Files/RADS/LI-RADS/LI-RADS-2018-Core.pdf?la=en
- See also: FACT-Hep questionnaire — https://www.facit.org/measures/FACT-Hep